CLINICAL TRIAL: NCT06773390
Title: Percutaneos Liver Biopsy in Pediatric Patient : Diagnostic Significance and Pattern of Liver Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohrail nagy naeim kerolos, Assiut government, Assiut University
Other Study IDs: Percutaneos liver biopsy
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Liver Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Percutaneous liver biposy — Percutaneous liver biopsy in pediatric patient diagnostic significance and pattern of liver diseases

SUMMARY:
In this study, we aim to evaluate the spectrum and pattern of liver diseases diagnosed by percutaneous tru-cut needle liver biopsy.

DETAILED DESCRIPTION:
Liver disease has a wide varied range of diseases that affect liver. In pediatrics, liver diseases can be categorized according to the underlying cause into: Acquired liver disease (as viral hepatitis, non-viral hepatitis, fatty liver, etc.), Autoimmune liver disease (Type1 autoimmune hepatitis, type 2 autoimmune hepatitis; thats more common in pediatrics), Congenital anomalies (biliary atresia, biliary (choledochal) cyst, Alagille syndrome), Metabolic liver disorder, a group of diseases occur when there is an abnormal gene in the metabolic pathway resulting in affection of the enzyme function, structure or amount, and Genetic diseases of liver (as Alpha 1 Antitrypsin Deficiency thats the most common genetic cause of liver disease in children) (1). However, liver disease may be part of a syndrome. In general, liver diseases are often asymptomatic in children; however commonest presenting signs and symptoms include jaundice, vomiting, coagulopathy or hepatomegaly (2,3).

In neonates, the first week of life is the mean age of onset of biliary atresia and galactosemia; however, symptoms may present in infancy. Also, viral hepatitis is commonly asymptomatic in neonates. In case of infants and children below 5 years, they may experience more presentation in liver disease. For example; glycogen storage diseases, alpha-1 antitrypsin deficiency, autoimmune hepatitis and others are more presented in the first five years of life. In neonates, infants and children; liver diseases are more common in males rather than females, except in autoimmune liver diseases; females are more common (2).

Diagnosis of liver disease in pediatrics represents a challenge because the majority of pediatrics has no symptoms especially in the early stages. Diagnostic tools of liver disease vary between laboratory investigation as Complete blood count (CBC), Liver function test (LFT), Viral markers, etc., imaging as abdominal ultrasonography (US), abdominal Computed tomography (CT),magnetic resonance imaging (MRI) and / or liver biopsy (4).

Liver biopsy is considered the best diagnostic tool in multiple diseases of liver and help clinicians in decision making. There are several types of liver biopsy: Percutaneous Liver Biopsy (PLB): it is the less invasive and the frequent used modality that can be conducted through physical examination (percussion over the upper right quadrant of the abdomen) or by sonar guidance. Trans-jugular Liver Biopsy; this technique is performed when patient has severe liver disease and coagulopathies or haematological condition and PLB is contraindicated. Surgical or Laparoscopic Liver biopsy; although it provides a large specimen size, it is done when there is increased risk of bleeding or in ascites of unknown cause and according to European Society for Pediatric Gastroenterology Hepatology and Nutrition

(ESPGHAN) laparoscopic liver biopsy used after failure of previous PLB, evaluation of abdominal mass or large liver sample for enzymatic analysis (5).

ELIGIBILITY:
Inclusion Criteria:

* All liver biopsy reports taken from infants and children with suspected liver disease aged less than 18 years between January 2019 and December 2023 who had been admitted in Pediatric Gastroenterology and Hepatology unit, Assiut University Children Hospital will be reviewed and included in the study.

Exclusion Criteria:

* Patients more than 18 years of age. Children with suspected Wilson Disease due to non-availability of the special stains used for histological diagnosis of the disease.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients aged less than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Identification of different patterns of liver diseases (inflammatory, metabolic, biliary abnormalities, cystic diseases of liver, others) and its correlation with clinical presentation. | Baseline

IPD SHARING:
Plan to Share IPD: No